CLINICAL TRIAL: NCT06482853
Title: Cardiovascular Effects of Angiotensin-(1-7) in Obesity Hypertension
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Amy Arnold, Associate Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY 8170-Part 2; R01HL170140 (NIH)
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Hypertension
Keywords: Angiotensin-(1-7); Cardiovascular; Sympathetic Nervous System; Blood Pressure; Endothelial Function
MeSH Terms: conditions — Obesity; Hypertension | interventions — angiotensin I (1-7); Acetates; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Angiotensin-(1-7) (Experimental): Participants will receive intravenous angiotensin-(1-7) at one study visit for a total of 120 minutes. Angiotensin-(1-7) will be given in escalating doses of 2 ng/kg/min, 4 ng/kg/min, and 8 ng/kg/min. Each of these doses will be infused for 10 minutes. Following this 30 minute dose escalation period, angiotensin-(1-7) will be given at 8 ng/kg/min for an additional 90 minutes. Infusion rates will be calculated for each patient based on body mass.
  Interventions: Drug: Angiotensin-(1-7)
- Saline (Placebo Comparator): Participants receive intravenous saline at one study visit for a total of 120 minutes. The volume of saline will match the volume of angiotensin-(1-7) infused. Infusion rates will be calculated for each patient based on body mass.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Angiotensin-(1-7) — This is a biologically active endogenous angiotensin peptide that may play an important role in regulation of blood pressure.
  Other Names: Angiotensin I/II (1-7) Acetate
  Arms: Angiotensin-(1-7)
Drug: Saline — Saline will be used as the placebo comparator.
  Other Names: Normal saline; 0.9% sodium chloride
  Arms: Saline

SUMMARY:
Obesity is a global health concern that is associated with high blood pressure and an increased risk for developing cardiovascular disease. The purpose of this study is to find out if the investigational drug angiotensin-(1-7) can improve cardiovascular health in people with obesity and high blood pressure.

DETAILED DESCRIPTION:
A randomized, double blind, placebo controlled, crossover study will be conducted to determine if acute intravenous angiotensin-(1-7) infusion reduces cardiovascular sympathetic tone and blood pressure and improves the function of blood vessels in participants with obesity hypertension. This is an outpatient study that requires a screening visit, and if eligible, two study visits separated by at least one week in the Clinical Research Center within the Penn State Milton S. Hershey Medical Center. The study visits will include intravenous infusion of angiotensin-(1-7) or saline for approximately two hours, starting with increasing doses and holding at a steady-state dose. Endothelial function will be measured and blood samples collected at baseline and at the end of infusion. Blood pressure, heart rate, and muscle sympathetic nerve activity (via microneurography) will be measured continuously throughout the study. Each study visit will last approximately 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all races
* Age 18 to 65 years
* Body mass index (BMI) between 30-45 kg/m2
* Pre-hypertension (defined as two or more seated blood pressure readings >120/80 mmHg) or hypertension (defined as two or more seated blood pressure readings >130/80 mmHg or use of antihypertensive medications)
* Capable of giving informed consent
* Fluent in written and spoken English
* Satisfactory history and physical exam

Exclusion Criteria:

* Age ≤ 17 or ≥ 66 years
* Taking more than two antihypertensive medications
* Secondary causes of hypertension (e.g., pheochromocytoma, primary aldosteronism, aortic coarctation, adrenal disease)
* Pregnant or nursing women
* Women taking hormone replacement therapy within 6 months
* Decisional impairment
* Prisoners
* Alcohol or drug abuse
* Current smokers
* Highly trained athletes
* Subjects with >5% weight change in the past 3 months
* BMI > 45 kg/m2
* Evidence of type I or type II diabetes (fasting glucose > 126 mg/dL or use of anti-diabetic medications)
* History of serious cardiovascular disease (e.g. myocardial infarction within 6 months, symptomatic coronary artery disease, presence of angina pectoris, significant arrhythmia, congestive heart failure, deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis, hypertrophic cardiomyopathy) or cerebrovascular disease (e.g. cerebral hemorrhage, stroke, transient Ischemic attack)
* History or presence of immunological or hematological disorders
* Impaired hepatic function [aspartate aminotransferase (AST) or alanine transaminase (ALT) levels >2 times upper limit of normal range]
* Impaired renal function (serum creatinine >2.0 mg/dl)
* Anemia
* Treatment with drugs increasing sympathetic activity [e.g., serotonin-norepinephrine reuptake inhibitors (SNRIs) or norepinephrine transporter (NET) inhibitors, stimulants]
* Treatment with phosphodiesterase-5 inhibitors
* Treatment with anticoagulants (e.g. warfarin)
* Treatment with chronic systemic glucocorticoid therapy (>7 consecutive days in 1 month)
* Treatment with any investigational drug in the 1-month preceding the study
* Inability to give, or withdraw, informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle Sympathetic Nerve Burst Rate | 120 minutes
  Muscle sympathetic nerve burst rate will be measured continuously using peroneal nerve microneurography during angiotensin-(1-7) versus saline infusion.
Change in Brachial Artery Diameter | 120 minutes
  A blood pressure cuff will be inflated to a suprasystolic pressure for 5 minutes then deflated. Brachial artery diameter will be measured continuously before, during, and after cuff inflation using duplex ultrasound at baseline and at the end of angiotensin-(1-7) versus saline infusion.

SECONDARY OUTCOMES:
Change in Muscle Sympathetic Nerve Burst Incidence | 120 minutes
  Muscle sympathetic nerve burst incidence will be measured continuously using peroneal nerve microneurography during angiotensin-(1-7) versus saline infusion.
Change in Muscle Sympathetic Nerve Amplitude | 120 minutes
  Muscle sympathetic nerve amplitude will be measured continuously using peroneal nerve microneurography during angiotensin-(1-7) versus saline infusion.
Change in Muscle Sympathetic Nerve Total Activity | 120 minutes
  Muscle sympathetic nerve total activity will be measured continuously using peroneal nerve microneurography during angiotensin-(1-7) versus saline infusion.
Change in Systolic Blood Pressure | 120 minutes
  Blood pressure will be measured continuously with a finger and arm cuff during angiotensin-(1-7) versus saline infusion.
Change in Diastolic Blood Pressure | 120 minutes
  Blood pressure will be measured continuously with a finger and arm cuff during angiotensin-(1-7) versus saline infusion.
Change in Heart Rate | 120 minutes
  Heart rate will be measured continuously by electrocardiogram during angiotensin-(1-7) versus saline infusion.
Change in Plasma Catecholamines | 120 minutes
  Circulating catecholamine levels will be measured in blood samples obtained at baseline and at the end of angiotensin-(1-7) versus saline infusion.

OTHER OUTCOMES:
Change in Angiotensin II | 120 minutes
  Plasma angiotensin II levels will be measured in blood samples obtained at baseline and at the end of angiotensin-(1-7) versus saline infusion.
Change in Angiotensin-(1-7) | 120 minutes
  Plasma angiotensin-(1-7) levels will be measured in blood samples obtained at baseline and at the end of angiotensin-(1-7) versus saline infusion.
Change in Renin Activity | 120 minutes
  Plasma renin activity will be measured in blood samples obtained at baseline and at the end of angiotensin-(1-7) versus saline infusion.
Change in Aldosterone | 120 minutes
  Plasma or serum aldosterone levels will be measured in blood samples obtained at baseline and at the end of angiotensin-(1-7) versus saline infusion.
Change in Heart Rate Variability | 120 minutes
  Heart rate variability will be calculated from the continuous electrocardiogram recordings obtained during angiotensin-(1-7) versus saline infusion.
Change in Baroreflex Sensitivity | 120 minutes
  Baroreflex sensitivity will be calculated from the continuous blood pressure and electrocardiogram recordings obtained during angiotensin-(1-7) versus saline infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Arnold, PhD, Principal Investigator — Pennsylvania State University College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.